CLINICAL TRIAL: NCT05232214
Title: Comparison of Three Swept-source Optical Coherence Biometry Devices in Long and Short Eyes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prof. Dr, Head of Department, Vienna Institute for Research in Ocular Surgery
Other Study IDs: Argos
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Cataract
Keywords: biometry
MeSH Terms: conditions — Cataract | interventions — Biometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- short eyes: Axial length under 22.5 mm
  Interventions: Device: Biometry
- long eyes: Axial length under 25.5 mm
  Interventions: Device: Biometry

INTERVENTIONS:
Device: Biometry — Only one eye from each patient will be included in the study. All patients included in the study will undergo biometric measurements in a random fashion with the three devices (IOLMaster 700, Argos and Anterion Heildelberg). Each patient will be measured three times with each device

SUMMARY:
The aim of the study is to compare the agreement and repeatability of ocular biometric parameters obtained using three swept-source optical coherence tomography (ss-OCT) device (Argos, IOLMaster 700 and ANTERION).

This is a prospective, single centre study, that would include a number of 50 eyes of 50 patients, which attend pre-surgical examination. Three measurements per biometry device will be performed on the day of the first eye surgery. The measurements will be performed in a randomised fashion with three ss-OCT devices (IOLMaster 700, Argos and ANTERION).

Inclusion criteria are: 40 years or above, age-related cataract, 20 eyes with AL< 22.0 mm and 30 eyes with AL>25.5 mm.

Exclusion criteria are: patients with ocular or systemic pathologies that would interfere with the measurements (e.g. dense cataract, corneal pathology, nystagmus).

The main outcome of the study will be: the difference (Limits of agreement) between the devices for the following parameters: keratometry (Ks, Kf, Km), CCT (µm), ACD (mm), LT (mm), AL (mm). Secondary outcomes will be: repeatability coefficient and coefficient of variation between the three device, measurement time for each device, and the feasibility for the Argos device.

DETAILED DESCRIPTION:
Accurate and repeatable biometric measurements are essential in providing an optimal refractive outcome.

ss-OCT biometry uses a tunable wavelength laser source to scan the eye, this technology showing its superiority through better signal-to-noise ratio, the wavelength light source being projected into the eye, one at a time; thus improving tissue penetration.

A previous study reported that the AL differs between adults was due mainly to the difference in vitreous cavity. The longer the AL becomes, the longer the posterior vitreous body becomes and the Argos defines the vitreous refractive index as 1.336. Therefore it is possible that the equivalent refractive index used in the IOLMaster 700 exceeds 1.336. Omoto et al. showed that the comparison of the arithmetic prediction errors between the Argos and IOLMaster 700 indicated that both biometers showed a myopic trend and the median arithmetic prediction errors were closer to zero with the Argos, the longer the AL became, this trend became more marked, suggesting that the Argos showed a significant hyperopic trend, especially with longer ALs.

This might show the advantage of using segmental refractive index instead of equivalent refractive index in longer ALs. Nevertheless, the authors did not include short eyes (<22mm) and longer AL (>32mm), thus further studies should be needed.

The aim of the study is to compare the agreement and repeatability of AL measurement using three different ssOCT devices in short (<22.5mm) and long eyes (>25.5mm).

This a prospective, randomised, observational study that would include patients (42 eyes of 42 patients) which attended pre-surgical examination. A written informed consent will be obtained from each patient.

Only one eye from each patient will be included in the study. All patients included in the study will undergo biometric measurements in a random fashion with the three devices (IOLMaster 700, Argos and Anterion Heildelberg). Each patient will be measured three times with each device and between the measurements they will be asked to blink or keep their eyes closed for tear film recovery and to avoid fatigue. Scans that pass the quality requirement of each device will be taken for analysis.

The order in which the measurements will be performed (Anterion, IOLMaster 700 or Argos) will be randomised using randomised.org.

Patients will be measured 8 weeks (+/-2 weeks) postoperatively with the three devices and the postoperative examination will also contain visual acuity, autorefraction and subjective refraction.

Each patient will receive the same type of lens (standard IOL, Clareon, Alcon). Inclusion criteria

* Written informed consent
* 21 years old or above
* age-related cataract
* AL<22.5 mm or >25.5 mm (long or short eyes) Exclusion criteria
* patients with dense cataract (LOCS grading III) or mature cataract
* corneal pathology that would significantly influence biometric measurements
* nystagmus or pathologies that would affect patient fixation
* pregnancy- for women in reproductive age a pregnancy test will be performed.

  • Main outcome: Limits of agreement (1.96xSD) between the optical biometers for the AL (mm) data

  • Secondary outcomes:
* Subgroup analysis for the refractive outcome (SEQ) after 8 weeks (+/-2 weeks) in short (<22,5mm) and long eyes (>25,5mm).
* Limits of agreement (1.96xSD) between the optical biometers for the following variables: keratometry (Ks, Kf, Km), CCT (µm), ACD (mm), LT (mm),
* Duration (seconds) of measurement time and total time (including data entry)
* Evaluation of the Barrett (and Haigis formulae with the 3 devices (mean of actual vs. mean of predicted SEQ)
* Repeatability coefficient (within subject standard deviation - SD) and coefficient of variation between the three devices

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 21 years old or above
* age-related cataract
* AL<22.5 mm or >25.5 mm (long or short eyes)

Exclusion Criteria:

* patients with dense cataract (LOCS grading III) or mature cataract
* corneal pathology that would significantly influence biometric measurements
* nystagmus or pathologies that would affect patient fixation
* pregnancy- for women in reproductive age a pregnancy test will be performed.

Ages: 21 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: age related cataract
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Axial length | 8Weeks
  Limits of agreement (1.96xSD) between the optical biometers for the AL (mm) data

SECONDARY OUTCOMES:
other Biometry parameter | 8 weeks
  - Limits of agreement (1.96xSD) between the optical biometers for the following variables: keratometry (Ks, Kf, Km), CCT (µm), ACD (mm), LT (mm),
Repeatability | 8 weeks
  - Repeatability coefficient (within subject standard deviation - SD) and coefficient of variation between the three devices

CONTACTS AND LOCATIONS:
Locations (1):
- Hanusch Hospital, Department of Ophthalmology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
All results will be shared in a published paper